CLINICAL TRIAL: NCT05993325
Title: A Phase III Multinational, Multicenter, Observer-Blinded, Randomized, Active-Controlled Trial to Evaluate the Immunogenicity and Safety of the Preventive COVID-19 Vaccine AdCLD-CoV19-1 OMI Administered As a Booster to Adults Aged 19 Years Old and Above
Brief Title: Immunogenicity and Safety of AdCLD-CoV19-1 OMI As a Booster: a COVID-19 Preventive Vaccine in Healthy Volunteers
Acronym: COVID-19
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COVENT-202
Record Dates: First submitted 2023-08-14; First posted 2023-08-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Vaccines
Keywords: COVID-19; SARS-CoV-2; Omicron; B.1.1.529
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 dose of AdCLD-CoV19-1 OMI (Experimental): Test group will receive 1 dose of AdCLD-CoV19-1 OMI
  Interventions: Biological: AdCLD-CoV19-1 OMI
- 1 dose of Comirnaty Bivalent (Active Comparator): Control group will receive 1 dose of Comirnaty Bivalent
  Interventions: Biological: Comirnaty Bivalent 0.1mg/mL (tozinameran and riltozinameran)

INTERVENTIONS:
Biological: AdCLD-CoV19-1 OMI — 3000 participants will receive investigational product (AdCLD-CoV19-1 OMI) via intramuscular administration in the deltoid muscle
  Arms: 1 dose of AdCLD-CoV19-1 OMI
Biological: Comirnaty Bivalent 0.1mg/mL (tozinameran and riltozinameran) — 1000 participants will receive investigational product (Comirnaty Bivalent) via intramuscular administration in the deltoid muscle
  Arms: 1 dose of Comirnaty Bivalent

SUMMARY:
The immunogenicity and safety of AdCLD-CoV19-1 OMI (5.0x10^10 VP (0.5 mL)/dose/Vial) administered as a booster in healthy adults aged 19 years old and above will be evaluated. Outcome assessment will be performed in comparison with Comirnaty Bivalent.

ELIGIBILITY:
Inclusion Criteria:

1. Individual aged 19 and above and willing to provide written informed consent to participate study voluntarily.
2. Individual fall under one or more of the following at the date of IP administration

   * At least past 16 weeks (112 days) without additional COVID-19 vaccination since the last COVID-19 vaccination.
   * At least past 16 weeks (112 days) since the release of quarantine due to COVID-19 confirmation.
3. Individual who agrees to use medically acceptable contraceptive methods† for at least 4 weeks prior to screening and 12 weeks post IP administration.
4. Individual who agrees not to donate or transfuse blood (including whole blood, plasma components, platelet components, platelet plasma components) throughout the study participation.

Exclusion Criteria:

1. Individual fall under one or more of the following at the date of IP administration

   * History of COVID-19 within 16 weeks (-111~0 days) or considered to be infected prior to IP administration.
   * History of receiving COVID-19 vaccine within 16 weeks (-111~0 days) prior to IP administration.
2. Clinically significant abnormalities on clinical laboratory tests, electrocardiograms, and chest X-rays performed during screening visit.
3. Positive HIV test result on the screening test.
4. Acute febrile illness with (≥38°C), or any suspected infectious diseases, or COVID-19-like symptoms (cough, shortness of breath, chills, myalgia, headache, sore throat, loss of taste/smell, etc.) within 3 days prior to administration of IP.
5. Any serious medical or psychiatric disease which in opinion of investigator judges unable to participate.

   * Respiratory diseases: Asthma, Chronic Obstructive Pulmonary Disease (COPD), active or latent tuberculosis which require medication, or individual who has received treatment due to worsening of the listed respiratory disease within 5 years prior to administration of IP.
   * Serious cardiovascular diseases: Congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension, thrombocytopenia or venous thrombosis, capillary leakage syndrome, myocarditis, pericarditis, etc.
   * Neurologic diseases: Epilepsy, seizure within past 3 years, migraine, stroke, encephalopathy, Guillain-Barre Syndrome, encephalomyelitis, transverse myelitis, etc.
   * Malignant cancer diagnosed within past 5 years (skin basal cell and squamous cell carcinoma are excluded).
   * Immune function disorders including autoimmune hypothyroidism, psoriasis.
   * Immunodeficiency diseases.
   * History of dependently administering psychotropic drugs or narcotic analgesics within 24 weeks prior to administration of IP, or psychiatric disease or behavioral impairment that, in the opinion of the investigator, could interfere with the participant's ability to participate in the study.
   * Other hepatobiliary, renal, endocrine, urinary tract, muscular skeletal diseases which the investigator considers clinically significant.
6. History of splenectomy.
7. Known history of allergic or hypersensitivity to the components of IP.
8. Known history of serious adverse reaction, allergies or hypersensitivity related to vaccination.
9. Individual with history of bleeding diathesis or thrombocytopenia, or history of severe bleeding or bruising after intramuscular injection or venipuncture or is receiving an anticoagulant (Individual receiving low dose aspirin (less than 100mg/day) can be enrolled in judgement of investigator).
10. History of hereditary or idiopathic angioneurotic edema.
11. History of systemic urticaria within 5 years prior to administration of IP.
12. Individual with history of solid organ or bone marrow transplantation.
13. Individual who is suspected or with history of drug or alcohol abuse within 24 weeks prior to administration of IP.
14. History of licensed drug for COVID-19 prevention aside from COVID-19 vaccine within 52 weeks prior to administration of IP.
15. Use of immunosuppressive or chronic use of systemic steroids within 6 weeks prior to administration of IP (Topical steroids, nasal spray and inhalers are allowed).

    * Immunosuppressive: Azathioprine, Cyclosporine, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, Cyclophosphamide, 6-Mercaptopurine, Methotrexate, Rapamycin, Leflunomide, etc.
    * Chronic steroid: >10 mg/day prednisone equivalent for periods exceeding 14 days.
16. Individual who has administered other investigational product or device within 24 weeks prior to screening visit.
17. Individual who has received or planned to receive any other vaccines within 28 days prior and after the administration of IP (Flu vaccines can be administered up to 14 days prior to the date of IP administration).
18. Receipt of immunoglobulin or blood-derived products within 12 weeks prior to administration of IP.
19. Individual with scheduled surgery throughout the study period.
20. Pregnant or lactating women.
21. Individual directly related to the investigator and meets the following:

    * Personnel relationship or subordinate-superior relationship (employees of the investigator's department, staffs of this trial).
    * Students or researchers in the immediate department of the school to which the investigator belongs (e.g., medical university).
22. Individual who is unfit for this study for any other reason in judgement of investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Ratio of GMT of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration | At 28 days post IP administration
  Ratio of GMT of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration (GMT of AdCLD-CoV19-1 OMI / GMT of Comirnaty Bivalent).
  Geometric mean titer (GMT): The value of multiplying the antibody titer of all available subjects (N) and take the Nth order root value.
Difference in seroresponse rate (SRR) of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration | At 28 days post IP administration
  Difference in seroresponse rate (SRR) of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration (SRR of AdCLD-CoV19-1 OMI - SRR of Comirnaty Bivalent).
  Seroresponse rate (SRR): Proportion of subjects whose antibody titer rise at least 4-fold at the measurement point compared to baseline. The titer is defined as half of detection limit if the titer before administration is below detection limit.

SECONDARY OUTCOMES:
SRR (proportion of subject who achieved seroresponse), GMT, GMFR of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 26, 52 weeks post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration. | At 26, 52 weeks post IP administration
  SRR (proportion of subject who achieved seroresponse), GMT (Geometric mean titer), GMFR (Ratio of GMT or GMC rise at the measurement point compared to baseline) of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 26, 52 weeks post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration.
Differences in SRR, GMT, GMFR of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration by serostatus of SARS-CoV-2 N protein antibody. | At 28 days post IP administration
  Differences in seroresponse rate (SRR), geometric mean titer (GMT), geometric mean fold rise (GMFR) of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration by serostatus of SARS-CoV-2 N protein antibody.
Differences in SRR, GMT, GMFR of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration by country. | At 28 days post IP administration
  Differences in seroresponse rate (SRR), geometric mean titer (GMT), geometric mean fold rise (GMFR) of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration by country.
Proportion of immediate adverse events (AE) | Within 30 minutes post IP administraiton
  Immediate adverse events occurred within 30 minutes (2 hours for ≥75 years old) post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration.
Proportion of solicited local and systemic AE | Within 7 days (Days 0 - 6) post IP administration
  Solicited AEs occurred within 7 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration.
Proportion of unsolicited AE | Within 28 days (Days 0 - 27) post IP administration
  Unsolicited AEs occurred within 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration.
Proportion of SAE | Throughout the study duration, 12 months post IP administration
Proportion of Adverse Event Of Special Interest (AESI) | Throughout the study duration, 12 months post IP administration
Proportion of Medically-Attended Adverse Events (MAAE) | Throughout the study duration, 12 months post IP administration
Proportion of clinically significant changes in clinical laboratory tests | At 28 days post IP administration
Proportion of clinically significant changes in vital signs | At 28 days post IP administration
Proportion of clinically significant changes in physical examination | At 28 days post IP administration

OTHER OUTCOMES:
SRR, GMT, GMFR of SARS-CoV-2 Wuhan strain and Variants of concern (VOC) neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration. | At 28 days post IP administration
SRR, GMT, GMFR of SARS-CoV-2 B.1.1.529 S protein-specific antibody measured by ELISA at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration. | At 28 days post IP administration
Cellular immune response (CMI) measured by ELISpot at 28 days, 26, 52 weeks post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration. | At 28 days, 26, 52 weeks post IP administration.
  Cellular immune response (CMI: responder rate, spot-forming unit) measured by ELISpot at 28 days, 26, 52 weeks post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration.
Differences of SRR, GMT, GMFR of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration by previous COVID-19 vaccination series. | At 28 days post IP administration
Differences of SRR, GMT, GMFR of SARS-CoV-2 B.1.1.529 neutralizing antibody measured by wild-type virus neutralization assay at 28 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration by age. | At 28 days post IP administration
Proportion of COVID-19 cases confirmed by antigen test from 14 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration to the end of the study. | Throughout the study duration, 12 months post IP administration
Proportion of severe COVID-19 cases from 14 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration to the end of the study. | Throughout the study duration, 12 months post IP administration
Proportion of hospitalization due to COVID-19 cases from 14 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration to the end of the study. | Throughout the study duration, 12 months post IP administration
Proportion of mortality due to COVID-19 cases from 14 days post AdCLD-CoV19-1 OMI or Comirnaty Bivalent administration to the end of the study. | Throughout the study duration, 12 months post IP administration

CONTACTS AND LOCATIONS:
Locations (17):
- Philippines (4):
  - The Medical City-Iloilo, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Tropical Disease Foundation, Inc., Makati
  - Far Eastern University - Nicanor Reyes Medical Foundation, Quezon City
- South Korea (13):
  - Dong-a University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - The Catholic University of Korea, ST. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Veterans Health Service Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No